CLINICAL TRIAL: NCT05393310
Title: Effects of Post Isometric Relaxation Versus Mulligan Mobilization With Movement on Pain, Disability and Dynamic Balance in Athletes With Chronic Ankle Sprain
Brief Title: Effects of MET vs Mulligan MWM on Pain, Disability & Balance in Athletes With Ankle Sprain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/22/0401 Faiz Ali
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Chronic Ankle Sprain
Keywords: ankle sprain, mulligan MWM, METs
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- post-isometric relaxation (Experimental): effects of post-isometric relaxation on pain, disability and dynamic balance in athletes with chronic ankle sprain
  Interventions: Other: post isometric relaxation
- mulligan mobilization with movement (Experimental): effects of mulligan mobilization with movement on pain, disability and dynamic balance in athletes with chronic ankle sprain
  Interventions: Other: MWM group

INTERVENTIONS:
Other: post isometric relaxation — The therapist will apply Post isometric relaxation ensure that foot will not actually move and only a static muscle contraction apply and held for 20 seconds. This will be followed by 2-3 second of relaxation, and then the foot passively stretched to dorsiflexion up to the palpated barrier and/or tolerance to stretch. This will continue until no further gains achieved 2 sets of 5 repetitions a day for 3 days a week for 4 weeks
  Arms: post-isometric relaxation
Other: MWM group — MWM group will receive inferior tibiofibular, talocrural, or cubometatarsal MWM 2-8 treatment sessions over 4 weeks.
  Arms: mulligan mobilization with movement

SUMMARY:
Ankle Sprains are the most common injury in Athletes and have a high rate of recurrence, pain, dynamic balance and disability is the leading cause of season break in athletes with chronic ankle sprain so as we see post isometric relaxation and Mulligan MWM are the useful techniques used to minimize pain, improve dynamic balance and to restrain athlete from disability due to chronic ankle sprain.

This study will be a randomized clinical trial,non probability convenience sampling technique will be used to collect the data. The sample size of athletes will be taken in this study to find the effect of post isometric relaxation and mulligan mobilization with movement in athletes.

DETAILED DESCRIPTION:
Ankle Sprains are the most common injury in Athletes and have a high rate of recurrence, pain, dynamic balance and disability is the leading cause of season break in athletes with chronic ankle sprain so as we see post isometric relaxation and Mulligan MWM are the useful techniques used to minimize pain, improve dynamic balance and to restrain athlete from disability due to chronic ankle sprain. As the effect of post isometric relaxation in comparison with Mulligan MWM has never been investigated in Athletes, the aim of this study is to investigate and compare the effect of these two techniques on athletes with chronic ankle sprain presented with pain, dynamic imbalance that leads to disability.

This study will be a randomized clinical trial and will be conducted in Pakistan sports board and Multan sports complex. The study will be completed within the time duration of six months. Non probability convenience sampling technique will be used to collect the data. The sample size of athletes will be taken in this study to find the effect of post isometric relaxation and mulligan mobilization with movement in athletes of PSB and MSC, aged 20-35 years, were allocated to both intervention group. The participants will be divided into two groups i-e, MET group and MWM group. MET group will receive post-isometric relaxation technique for gastrocnemius and soleus muscle. Patient will be in prone lying with the ankle out of the bed. 30% of the available strength will applied by the patient against unyielding resistance towards plantarflexion. The therapist will ensure that foot will not actually move and only a static muscle contraction apply and held for 20 seconds. This will be followed by 2-3 second of relaxation, and then the foot passively stretched to dorsiflexion up to the palpated barrier and/or tolerance to stretch. This will continue until no further gains achieved 2 sets of 5 repetitions a day for 3 days a week for 4 weeks. MWM group will receive inferior tibiofibular, talocrural, or cubometatarsal MWM 2-8 treatment sessions over 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of chronic ankle sprain (grade I or II) (3-4 months)
* Players have spent at least one year in sports

Exclusion Criteria:

* • Players undergone surgery or had an accident.

  * Any malignant or chronic disease
  * Players with the history of fracture in the same ankle

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4th week
  Changes from baseline numeric pain rating scale for pain from 0-10 (0 means no pain and 10 means worst pain)
Dorsiflexion lunge test | 4th week
  Participants are instructed to lunge forward until their knee touches the wall (vertical line). The heel is required to remain in contact with the floor at all times. The foot is moved away from the wall to the point where the knee can only make slight contact with the wall, while the heel remains in contact with the floor. This puts the ankle joint in maximal dorsiflexion. The leg not being tested can rest on the the floor and participants are allowed to hold onto the wall for support. The maximum distance from the wall to the tip of the big toe is recorded. The distance is measured in centimeters (cm) with each centimeter corresponding to approximately 3.6° of ankle dorsiflexion
star excursion balance test | 4th week
  The Star Excursion Balance Test is a dynamic test that requires strength, flexibility, and proprioception.
Foot and Ankle outcome score | 4th week
  ankle disability

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Pakistan sports board, Lahore, Punjab Province
  - PSB, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hertel J. Functional Anatomy, Pathomechanics, and Pathophysiology of Lateral Ankle Instability. J Athl Train. 2002 Dec;37(4):364-375. PMID 12937557
- [Background] McGovern RP, Martin RL. Managing ankle ligament sprains and tears: current opinion. Open Access J Sports Med. 2016 Mar 2;7:33-42. doi: 10.2147/OAJSM.S72334. eCollection 2016. PMID 27042147
- [Background] Mohd Salim NS, Umar MA, Shaharudin S. Effects of the standard physiotherapy programme on pain and isokinetic ankle strength in individuals with grade I ankle sprain. J Taibah Univ Med Sci. 2018 Nov 30;13(6):576-581. doi: 10.1016/j.jtumed.2018.10.007. eCollection 2018 Dec. PMID 31435381
- [Background] Doherty C, Bleakley C, Hertel J, Caulfield B, Ryan J, Delahunt E. Dynamic balance deficits in individuals with chronic ankle instability compared to ankle sprain copers 1 year after a first-time lateral ankle sprain injury. Knee Surg Sports Traumatol Arthrosc. 2016 Apr;24(4):1086-95. doi: 10.1007/s00167-015-3744-z. Epub 2015 Aug 8. PMID 26254090
- [Background] Golightly YM, Devellis RF, Nelson AE, Hannan MT, Lohmander LS, Renner JB, Jordan JM. Psychometric properties of the foot and ankle outcome score in a community-based study of adults with and without osteoarthritis. Arthritis Care Res (Hoboken). 2014 Mar;66(3):395-403. doi: 10.1002/acr.22162. PMID 24023029